CLINICAL TRIAL: NCT07303387
Title: An Open Label Phase II Platform Modular Study Exploring the Efficacy and Safety of the Valemetostat (EZH1/2 Inhibitor) in Patients With Selected Solid Tumors
Brief Title: Efficacy and Safety of the Valemetostat in Patients With Selected Solid Tumors.
Acronym: EZHiSWITCH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-519788-16-00; 2024/3993 (Other: CSET Number (Gustave Roussy ID))
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Malignancies; Clear Cell Endometrial Carcinoma; Ovarian Cancer
Keywords: solid tumor; chromatin remodeling deficiency; Valemetostat; EZH1/2 inhibitor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valemetostat treatment (Experimental): After confirmation by IHC of the loss of expression in tumors cells of SMARCB1, SMARCA4, SMARCA2, SMARCC1, SMARCC2, ARID1A, ARID1B, PBRM1, BAP1and other SWI/SNF sub-units patients will included in different cohorts depending of gene with loss of expression. They will be all treated by Valemetostat
  Interventions: Drug: Valemetostat Tosylate

INTERVENTIONS:
Drug: Valemetostat Tosylate — Experimental treatment with Valemetostat (200mg per day), divided into 28-day periods called treatment cycles, for a maximum of two years

SUMMARY:
Rational, objective and design: Some cancer-protecting genes are inactivated when the EZH2 enzyme is too active or the SWI/SNF complex is less active. The EZH1/2 enzymes and the SWI/SNFs complex play opposing roles in gene expression: we hypothesize that valemetostat, an inhibitor of the EZH1/2 enzymes, will stop/slow down the growth of cancer cells by reactivating these genes. Numerous clinical trials are currently underway worldwide to optimize the development of valemetostat tosylate and potentially offer a new targeted therapeutic option for patients suffering from various cancer pathologies.

The aim of this research is to evaluate the efficacy of valemetostat on solid tumors, which have an alteration in certain genes: SMARC (B1/A4/A2/C1/C2), ARID (1A/1B), PBRM1, BAP1 and other SWI/SNF sub-units. The research will be conducted in two phases: 1) Pre-selection of patients with the desired alterations. 2) Treatment with valemetostat, 200mg/day, for a maximum of 2 years, with examinations every 28 days.

This is a multicenter, international, phase II open-label, multicenter modular study exploring the efficacy and safety of valemetostat. Module 1 will be the SWI/SNF basket monotherapy study describe below. Such design will allow the study to evolve considering signals for further monotherapy and/or combination modules.

The Primary endpoint of the study is Overall Response Rate at 24 weeks, defined as the proportion of patients with a confirmed best overall response.

Trial population: Adult patients with histologically/cytologically confirmed progressive metastatic or recurrent solid tumor, who have selected chromatin remodeling deficiency in at least one of the following genes: SMARCB1, SMARCA4, SMARCA2, SMARCC1, SMARCC2, ARID1A, ARID1B, PBRM1, BAP1and other SWI/SNF sub-units; or molecularly (Wildtype) and phenotypically-selected Clear cell endometrial or ovarian carcinoma cancers. Patients must be using an effective method of contraception and have signed the consent form. They must not participate in another clinical study with an investigational product during the last 3 weeks, during the study treatment and not have a contraindication to the study treatment (…) Intervention: After confirmation by IHC of the loss of expression in tumors cells of SMARCB1, SMARCA4, SMARCA2, SMARCC1, SMARCC2, ARID1A, ARID1B, PBRM1, BAP1and other SWI/SNF sub-units and validation of inclusion/exclusion criteria patients will included in different cohorts (refer to investigation scheme). All patients will receive Valemetostat (200 mg per day), divided into 28-day periods called treatment cycles, for a maximum of two years. The main interventions scheduled are blood samples (to evaluate biological parameters and for translational research), electrocardiogram, echocardiography and CTscan. For patients who have consented, sequential biopsies will be performed as follow: at baseline, on treatment and at progression.

Ethical consideration: This research will make it possible to collectively evaluate the interest of EZH1/2 inhibitor in solids tumors with SWI/SNF defect. Individually, by participating in this research, patients could benefit from these treatments based on cell-based results and in the treatment of relapsed/refractory peripheral T-cell lymphomas, with an improvement in symptoms and quality of life. As with any research, the investigational drug and other procedures that take place may involve risks, some of which are already known and others not yet described. The main risks (described in the consent form) are side effects of the valemetostat. If they agree, patients will also be monitored more closely with their safety assessed through patient-reported outcomes (PRO), the evaluation of their experience through qualitative interviews & assessment of quality of care and the evaluation of their biometric physiological via a wearable device.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
2. Ability to comply with the protocol.
3. Age ≥ 18 years.
4. Patients must have histologically or cytologically confirmed progressive metastatic or recurrent solid tumor (as defined below for each tumor type). Diagnosis must be stated in a pathology report and confirmed by the investigator.
5. Evidence of disease progression prior to trial entry.
6. Have exhausted all other standard-of-care therapeutic options which have shown efficacy in their disease and are expected to be more effective than valemetostat based on current evidence for standard-of-care and EZH1/2 inhibitors
7. Have an archival tissue sample available with sufficient tumor tissue for IHC confirmation of loss expression (20 slides required). If patients do not have sufficient archival material, a new biopsy should be scheduled.
8. Have documented bi-allelic (homozygous) deletion of SMARCB1, SMARCA4/2, ARID1A/B, PBRM1, BAP1, SMARCC1/2 or other SWI/SNF in a tumor detected by a validated NGS test (solid or liquid) and confirmed loss of expression in tumour cells by centralized IHC.

   Cohort 1.A - SMARCB1-defective (maximum of 1 prior treatment line) Cohort 1.B - SMARCA4 (maximum of 3 prior treatment lines) Cohort 1.C - ARID1A (maximum of 2 prior treatment lines) Cohort 1Ca: Endometrial and ovarian clear cell only Cohort 1Cb: Other ARID1A-defective tumors Cohort 1.D - PBRM1 (with a minimum of 6 clear cell renal cell carcinoma during stage 1; maximum of 3 prior treatment lines) Cohort 1.E - BAP1 (with a maximum of 5 mesothelioma during stage 1; maximum of 2 prior treatment lines) Cohort 1.F - SMARCA2 or other SWI/SNF subunits (maximum of 2 prior treatment lines) Cohort 1.G - Clear cell Endometrial or Ovarian carcinoma SWI/SNF wild-type (maximum of 2 prior treatment lines) Tissue used for assessing SWI/SNF or BAP1 status must be < 3 years old; otherwise, a new fresh biopsy should be performed.
9. At least one lesion, not previously irradiated, measurable according to RECIST v1.1 (PCWG3/RECIST1.1 for prostate cancer and mRECIST for pleural mesothelioma) as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and suitable for repeated assessment.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration at the time of enrollment.
11. Estimated life expectancy of greater than 12 weeks.
12. Adequate hematologic and organ function, defined by the following laboratory results obtained within 3 days prior to the first study treatment (Cycle 1 Day 1):

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/μL (without granulocyte colony-stimulating factor support within 14 days prior to the screening assessment).
    2. Lymphocyte count ≥ 500/μL.
    3. Platelet count ≥ 100.000/μL (platelet transfusion is not allowed within 14 days prior to the screening assessment).
    4. Hemoglobin ≥ 9g/dL (packed red blood cell transfusion is not allowed within 14 days prior to the screening assessment).
    5. Total bilirubin ≤ 1.5 ULN (subjects with documented/suspected Gilbert's disease can have total bilirubin ≤3x ULN and direct bilirubin ≤1.5x ULN or subjects with liver metastases at baseline can have total bilirubin ≤ 3 × ULN).
    6. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤ 3.0x upper normal limit (ULN) or ≤ 5 × ULN in case of liver metastases.
    7. Albumin ≥ 2.5g/dL.
    8. Creatinine clearance ≥ 40 mL/min (according to Cockroft and Gault formula).
    9. International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular weight heparin or warfarin) should be on stable dose and must have PT-INR within therapeutic range as deemed appropriate by the Investigator.
13. Women of childbearing potential must have at least one negative serum β-HCG pregnancy test during the screening assessment. Prior to the administration of the first study treatment, there must be a negative serum β-HCG pregnancy test within 72 hours prior or a negative urine pregnancy test within 24 hours prior. Women of childbearing potential must have a negative serum pregnancy test at Screening and must be willing to use highly effective birth control, upon enrollment, during the Treatment Period, and for 3 months, following the last dose of study drug administration.

    A woman is considered of childbearing potential following menarche and until becoming post-menopausal (≥ 12 months of non-therapy-induced amenorrhea) unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral oophorectomy and bilateral salpingectomy with surgery at least 1 month before the first dose of study drug or confirmed by follicle stimulating hormone (FSH) test >40 mIU/mL and estradiol <40 pg/mL (<140 pmol/L).
14. Sexually active women of childbearing potential must agree to use a highly effective method of contraception << supplemented by a barrier method >>, or to abstain from sexual activity during the study and for at least 3 months after the last dose of study treatment.
15. Participant must agree to not breastfeed during the study or for 3 months after the last dose of study treatment.
16. Sexually active male's patients with partner of childbearing potential, the subject must be surgically sterile or willing to use highly effective birth control upon enrollment, during the Treatment Period, and for 3 months following the last dose of study drug.
17. Participant must agree to not donate blood during the study or for 3 months days after the last dose of study treatment.
18. Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and for at least 3 months after the final study drug administration.
19. Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 3 months after the final study drug administration.
20. Patient should be able and willing to comply with study visits and procedures as per protocol.
21. Patients must be affiliated to a social security system or beneficiary of an equivalent system.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 4 weeks (excepting observational or non-interventional clinical studies).
2. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 21 days prior to the first dose of study drug, or five half-lives of the previous agent, whichever is the longer.
3. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks prior to Cycle 1 Day 1; or curative radiation therapy or major surgery within 4 weeks or palliative radiation therapy within 2 weeks prior to Cycle 1 Day 1.
4. History of another primary malignancy within 5 years prior to Cycle 1 Day 1 except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease (eg, carcinoma in situ of the cervix, ductal carcinoma in situ treated surgically with curative intent).
5. Treatment with systemic (>10 mg daily prednisone equivalents). or other immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents) within 2 weeks prior to Cycle 1 Day 1, or anticipated requirements for systemic immunosuppressive medications during the trial:

   The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids for patients with orthostatic hypotension, low-dose supplemental corticosteroids for adrenocortical insufficiency and topical steroids for cutaneous diseases are allowed.
6. Acute toxicities from previous therapies that have not resolved to Grade ≤ 1, with the exception of alopecia.
7. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins. Known or suspected hypersensitivity to valemetostat tosylate or any of the excipients.
8. Uncontrolled or significant cardiovascular disease, including the following:

   1. Evidence of prolongation of QT/QTc interval (eg, repeated episodes of QT corrected for heart rate using Fridericia's method [QTcF] >470 ms) (average of triplicate determinations) refer to APPENDIX 9.
   2. Myocardial infarction within 6 months prior to Screening.
   3. Uncontrolled angina pectoris within 6 months prior to Screening.
   4. New York Heart Association (NYHA) Class 3 or 4 congestive heart failure.
   5. Uncontrolled hypertension (resting systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg).
   6. Patients with known left ventricular ejection fraction (LVEF) < 40%; patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable cardiologic treatment.
9. Known positive test for HIV or known acquired immunodeficiency syndrome
10. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection within 28 days prior to the first dose of study drug (hepatitis B surface antigen positive or have detectable HBV DNA or detectable HCV RNA).
11. Active tuberculosis.
12. Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection requiring treatment with intravenous antibiotics, antivirals, or antifungals. Note: Subjects with localized fungal infections of skin or nails are eligible.
13. Any active uncontrolled systemic diseases or other medical conditions considered to be poorly controlled by the investigator, including, but not limited to, bleeding diatheses
14. Current use of moderate or strong cytochrome P450 (CYP)3A inducers (Table 8)
15. Administration of attenuated or live vaccine within 4 weeks prior to Cycle 1 Day 1 or anticipation that such a live attenuated vaccine will be required during the study (except anti-COVID-19 vaccines).
16. Major surgical procedure within 20 days prior ty Cycle 1 Day 1 or anticipation of need for a major surgical procedure during the course of the study.
17. Uncontrolled tumor-related pain: patients requiring pain medication must be on a stable regimen at study entry and symptomatic lesions amenable to palliative radiotherapy should be treated prior to enrolment.
18. Uncontrolled effusion (pleural, pericardial or ascites) requiring recurrent drainage procedures (once a month or more frequently); patients with indwelling catheters (e.g. PleurX) are allowed.
19. Uncontrolled hypercalcemia (>1.5mmol/L ionized calcium or Ca > 12mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
20. History of leptomeningeal disease
21. Symptomatic CNS metastasis or uncontrolled CNS metastasis, requiring increasing doses of steroids or stable dose of steroids > 10mg prednisone QD.
22. Spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to Cycle 1 Day 1.
23. Female subjects who are pregnant, breast-feeding or male / female patients of reproductive potential who are not employing an effective method of birth control.
24. Previous treatment with EZH2 (or EZH1/2) inhibitors, except for cohort 1A where EZH2 inhibitors are approved.
25. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study result.
26. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2032-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the antitumor activity of valemetostat | From enrollment to visit at week 24
  Overall Response Rate defined as the proportion of patients with a confirmed best overall response of either CR or PR according to RECISTv1.1 (for all patients, except prostate), mRECIST v1.1 (mesothelioma), RECIST1.1/PCWG3 (prostate) and Choi Criteria (sarcoma)

SECONDARY OUTCOMES:
Ability of valemetostat to influence tumor growth | From enrollment to visit at week 24 and 12 months
  • Tumor Growth Rate (G-score)
Overall Survival | Through study completion, an average of 1 year
  • Overall survival (OS)
Incidence of AEs | Through study completion, an average of 1 year
  Incidence of AEs (including SAE and AESIs) according to the NCI CTCAE v5.0
Severity of AEs | Through study completion, an average of 1 year
  Severity of AEs (including SAE and AESIs) according to the NCI CTCAE v5.0
Disease Control Rate | From enrollment to visit at week 24 + Until the end of the study, an average of 1 year
Change in tumor size | From enrollment to visit at week 24 + Until the end of the study, an average of 1 year
  Percentage of change from baseline in tumor size
Duration Of Response | From enrollment to visit at week 24 + Until the end of the study, an average of 1 year
Best Overall Response Rate | From enrollment to visit at week 24 + Until the end of the study, an average of 1 year
Progression-free survival | From enrollment to visit at week 24 and 12 months
  PFS ratio on valemetostat (PFS pre-treatment / PFS on-treatment)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Gustave Roussy, Villejuif, Val de Marne
  - Institut Bergonié, Bordeaux
  - Centre Léon Berard, Lyon
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: No